CLINICAL TRIAL: NCT01738594
Title: A Randomized Phase I Dose-Escalation Trial of Carfilzomib With and Without Romidepsin in Cutaneous T-Cell Lymphoma
Brief Title: Dose-Escalation Trial of Carfilzomib With and Without Romidepsin in Cutaneous T-Cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Northwestern University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Barbara Pro, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 12H06; STU00071042 (Other: Northwestern University IRB); NCI-2012-01952 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2012-11-21; First posted 2012-11-30 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-04

CONDITIONS: Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IA Mycosis Fungoides/Sezary Syndrome; Stage IB Mycosis Fungoides/Sezary Syndrome; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IIA Mycosis Fungoides/Sezary Syndrome; Stage IIB Mycosis Fungoides/Sezary Syndrome; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IIIA Mycosis Fungoides/Sezary Syndrome; Stage IIIB Mycosis Fungoides/Sezary Syndrome; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IVA Mycosis Fungoides/Sezary Syndrome; Stage IVB Mycosis Fungoides/Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — carfilzomib; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (carfilzomib) (Experimental): Patients receive carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16.
  Interventions: Drug: carfilzomib; Other: laboratory biomarker analysis
- Arm B (carfilzomib, romidepsin) (Experimental): Patients receive carfilzomib as in Arm A and romidepsin IV over 4 hours on days 1, 8, and 15.
  Interventions: Drug: carfilzomib; Drug: romidepsin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax
  Arms: Arm B (carfilzomib, romidepsin)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I trial studies the side effects and the best dose of carfilzomib when given together with or without romidepsin in treating patients with stage IA-IVB cutaneous T-cell lymphoma. Carfilzomib and romidepsin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving carfilzomib alone is more effective than when given together with romidepsin.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of carfilzomib, both as a single agent as well as in combination with romidepsin, in patients with cutaneous T-cell lymphoma (CTCL).

SECONDARY OBJECTIVES:

I. Overall response rate (ORR). II. Duration of response. III. Time to progression (TTP).

TERTIARY OBJECTIVES:

I. Measure proteasome activity concurrently in peripheral blood mononuclear cells (PBMCs) and tumor tissue biopsy specimens in order to gather pilot data on proteasome inhibition in CTCL patients treated with carfilzomib alone as well as carfilzomib with romidepsin.

OUTLINE: This is a dose-escalation study of carfilzomib. Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive carfilzomib intravenously (IV) over 30 minutes on days 1, 2, 8, 9, 15, and 16.

ARM B: Patients receive carfilzomib as in Arm A and romidepsin IV over 4 hours on days 1, 8, and 15.

In both arms, treatment repeats every 28 days for at least 2-4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological confirmation of a cutaneous T-cell lymphoma (CTCL) of any histology; confirmation of histological diagnosis must be completed prior to enrollment by the lead site (Northwestern)

  * Patients will be stratified by mycosis fungoides (MF) and Sezary syndrome (SS) (report diagnostic or consistent with MF/SS), stage IA-IVB according to TNM blood (TNMB) classification versus other CTCL histologies
* Patients must have measurable disease (using modified Severity-Weighted Assessment Tool [mSWAT]) and/or use of indicator lesions must be designated prior to study enrollment (from imaging); measurable disease upon physical exam with a negative scan is acceptable
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients must have a life expectancy of >= 3 months
* Patients with MF/SS must have failed at least 1 prior topical therapy (including steroids, nitrogen mustard, retinoids, phototherapy, photochemotherapy, radiation, and total skin electron beam); there is no upper limit for prior therapies
* Serum creatinine =< 2.0 mg/dL
* Total bilirubin =< 2.2 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2 x upper limit of normal (ULN)
* Leukocytes >= 3,000/mm^3
* Absolute neutrophils >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Patients must have an electrocardiogram (EKG) demonstrating QTc =< 500 ms within 28 days prior to registration
* Females of child-bearing potential and sexually active males must agree to use effective methods of contraception:

  * Child-bearing potential is defined as any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has NOT undergone a hysterectomy or bilateral oophorectomy; OR
    * Has NOT been naturally menopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months)
  * The effectiveness of hormonal contraceptives may be reduced by romidepsin, thus effective methods should include at least 1 form of barrier contraception
* Females of child-bearing potential must have a negative pregnancy test within 7 days prior to registration
* Patients must be disease free of any prior malignancies for >= 3 years

  * The exception to this would be currently treated squamous cell and basal cell carcinoma of the skin, carcinoma in situ of the cervix, breast, or bladder, or surgically removed melanoma in situ of the skin (stage 0) with histologically confirmed free margins of excision
* Patients must give written informed consent prior to registration on the study

Exclusion Criteria:

* Patients who have received topical therapy, systemic chemotherapy, or biological therapy within 4 weeks prior to registration are NOT eligible for participation
* Patients who have undergone major surgery within 21 days prior to registration are NOT eligible for participation
* Patients who have an acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to registration are NOT eligible for participation
* Patients in whom IV fluid hydration is contraindicated (e.g. due to pre-existing pulmonary, cardiac, or renal impairment) will NOT be eligible for participation
* Patients who are pregnant and/or lactating are NOT eligible for participation
* Patients who have had a prior stem cell transplantation are NOT eligible for participation
* Patients who have had any of the following cardiac conditions are NOT eligible for participation (unless otherwise noted):

  * Unstable angina or myocardial infarction within 4 months prior to registration
  * New York Heart Association (NYHA) class II or IV heart failure
  * Uncontrolled angina
  * A history of severe coronary artery disease
  * Severe, uncontrolled ventricular arrhythmias
  * Sick sinus syndrome
  * Electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities UNLESS the patient has a pacemaker
* Patients who exhibit uncontrolled hypertension (>= 140/90 mmHg) or uncontrolled diabetes within 14 days prior to registration are NOT eligible for participation
* Patients who have experienced significant neuropathy (grades 3-4 or grade 2 with pain) within 14 days prior to registration are NOT eligible for participation
* Patients who have a known history of allergy to Captisol (a cyclodextrin derivative used to stabilize carfilzomib) are NOT eligible for participation
* Patients who have a contraindication to any of the required concomitant drugs or supportive treatments (including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment) are NOT eligible for participation
* Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to registration are NOT eligible for participation
* Patients who have any serious condition, laboratory abnormality, or psychiatric illness that would prevent them from singing the informed consent form are NOT eligible for participation
* Patients who have had prior exposure to romidepsin or any proteasome inhibitor are NOT eligible for participation
* Patients with a known human immunodeficiency virus (HIV) infection are NOT eligible for participation
* Patients who test positive for infectious hepatitis types A, B, or C within 14 days of registration are NOT eligible for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-03-22 (Actual); Primary Completion 2016-10-11 (Actual); Study Completion 2016-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pro, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on December 19, 2012 with the first patient being enrolled on March 22, 2013 and an accrual goal of up to 48 patients. The study was designed as a dose escalation with 3+3 cohorts and two arms. The study was closed to further accrual of patients on September 13, 2016 due to slow accrual.
Groups:
- Arm A, Cohort -1 (Carfilzomib): Patients receive carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16 of each 28 day cycle.
  Cycle 1 day 1 dose will be 20 mg/m2, all subsequent doses (of cycle 1 and future cycles) will be stepped up to 27 mg/m2.
  carfilzomib: Given IV
  laboratory biomarker analysis: Correlative studies
- Arm A, Cohort 1 (Carfilzomib): Patients receive carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16 of each 28 day cycle.
  Cycle 1 day 1 dose will be 20 mg/m2, all subsequent doses (of cycle 1 and future cycles) will be stepped up to 36 mg/m2.
  carfilzomib: Given IV
  laboratory biomarker analysis: Correlative studies
- Arm A, Cohort 2 (Carfilzomib): Patients receive carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16 of each 28 day cycle.
  Cycle 1 day 1 dose will be 20 mg/m2, all subsequent doses (of cycle 1 and future cycles) will be stepped up to 45 mg/m2.
  carfilzomib: Given IV
  laboratory biomarker analysis: Correlative studies
- Arm A, Cohort 3 (Carfilzomib): Patients receive carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16 of each 28 day cycle.
  Cycle 1 day 1 dose will be 20 mg/m2, all subsequent doses (of cycle 1 and future cycles) will be stepped up to 56 mg/m2.
  carfilzomib: Given IV
  laboratory biomarker analysis: Correlative studies
- Arm B Cohort -1 (Carfilzomib + Romidepsin): Patients receive carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16 of each 28 day cycle.
  Cycle 1 day 1 dose will be 20 mg/m2, all subsequent doses (of cycle 1 and future cycles) will be stepped up to 27 mg/m2.
  and romidepsin IV over 4 hours on days 1, 8, and 15 of each 28 day cycle.
  carfilzomib: Given IV
  romidepsin: Given IV
  laboratory biomarker analysis: Correlative studies
- Arm B Cohort 1 (Carfilzomib + Romidepsin: Patients receive carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16 of each 28 day cycle.
  Cycle 1 day 1 dose will be 20 mg/m2, all subsequent doses (of cycle 1 and future cycles) will be stepped up to 36 mg/m2.
  and romidepsin IV over 4 hours on days 1, 8, and 15 of each 28 day cycle.
  carfilzomib: Given IV
  romidepsin: Given IV
  laboratory biomarker analysis: Correlative studies
- Arm B Cohort 2 (Carfilzomib + Romidepsin): Patients receive carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16 of each 28 day cycle.
  Cycle 1 day 1 dose will be 20 mg/m2, all subsequent doses (of cycle 1 and future cycles) will be stepped up to 45 mg/m2.
  and romidepsin IV over 4 hours on days 1, 8, and 15 of each 28 day cycle.
  carfilzomib: Given IV
  romidepsin: Given IV
  laboratory biomarker analysis: Correlative studies
- Arm B Cohort 3 (Carfilzomib + Romidepsin): Patients receive carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16 of each 28 day cycle.
  Cycle 1 day 1 dose will be 20 mg/m2, all subsequent doses (of cycle 1 and future cycles) will be stepped up to 56 mg/m2.
  and romidepsin IV over 4 hours on days 1, 8, and 15 of each 28 day cycle.
  carfilzomib: Given IV
  romidepsin: Given IV
  laboratory biomarker analysis: Correlative studies
Period: Registration and Treatment Start
Arm/Group | Arm A, Cohort -1 (Carfilzomib) | Arm A, Cohort 1 (Carfilzomib) | Arm A, Cohort 2 (Carfilzomib) | Arm A, Cohort 3 (Carfilzomib) | Arm B Cohort -1 (Carfilzomib + Romidepsin) | Arm B Cohort 1 (Carfilzomib + Romidepsin | Arm B Cohort 2 (Carfilzomib + Romidepsin) | Arm B Cohort 3 (Carfilzomib + Romidepsin)
Started | 0 | 3 | 0 | 0 | 1 | 3 | 0 | 0
Registered to Study | 0 | 3 | 0 | 0 | 1 | 3 | 0 | 0
Treatment Started | 0 | 2 | 0 | 0 | 1 | 3 | 0 | 0
Completed | 0 | 2 | 0 | 0 | 1 | 3 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Completed 2 Cycles/Reached 1st Response
Arm/Group | Arm A, Cohort -1 (Carfilzomib) | Arm A, Cohort 1 (Carfilzomib) | Arm A, Cohort 2 (Carfilzomib) | Arm A, Cohort 3 (Carfilzomib) | Arm B Cohort -1 (Carfilzomib + Romidepsin) | Arm B Cohort 1 (Carfilzomib + Romidepsin | Arm B Cohort 2 (Carfilzomib + Romidepsin) | Arm B Cohort 3 (Carfilzomib + Romidepsin)
Started | 0 | 2 | 0 | 0 | 1 | 3 | 0 | 0
Completed | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Completed 4 Cycles of Treatment
Arm/Group | Arm A, Cohort -1 (Carfilzomib) | Arm A, Cohort 1 (Carfilzomib) | Arm A, Cohort 2 (Carfilzomib) | Arm A, Cohort 3 (Carfilzomib) | Arm B Cohort -1 (Carfilzomib + Romidepsin) | Arm B Cohort 1 (Carfilzomib + Romidepsin | Arm B Cohort 2 (Carfilzomib + Romidepsin) | Arm B Cohort 3 (Carfilzomib + Romidepsin)
Started | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not Completed | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive disease | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No response/patient benefit | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Went on to Continue Treatment Cycle 5
Arm/Group | Arm A, Cohort -1 (Carfilzomib) | Arm A, Cohort 1 (Carfilzomib) | Arm A, Cohort 2 (Carfilzomib) | Arm A, Cohort 3 (Carfilzomib) | Arm B Cohort -1 (Carfilzomib + Romidepsin) | Arm B Cohort 1 (Carfilzomib + Romidepsin | Arm B Cohort 2 (Carfilzomib + Romidepsin) | Arm B Cohort 3 (Carfilzomib + Romidepsin)
Started | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Follow up for 1 Year
Arm/Group | Arm A, Cohort -1 (Carfilzomib) | Arm A, Cohort 1 (Carfilzomib) | Arm A, Cohort 2 (Carfilzomib) | Arm A, Cohort 3 (Carfilzomib) | Arm B Cohort -1 (Carfilzomib + Romidepsin) | Arm B Cohort 1 (Carfilzomib + Romidepsin | Arm B Cohort 2 (Carfilzomib + Romidepsin) | Arm B Cohort 3 (Carfilzomib + Romidepsin)
Started (All patients that receive treatment on study go into the follow up period) | 0 | 2 | 0 | 0 | 1 | 3 | 0 | 0
Completed | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Some arms did not accrue patients due to the study closing for slow accrual.
Groups:
- Arm B Cohort 1 (Carfilzomib + Romidepsin): Patients receive carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16 of each 28 day cycle.
  Cycle 1 day 1 dose will be 20 mg/m2, all subsequent doses (of cycle 1 and future cycles) will be stepped up to 36 mg/m2.
  and romidepsin IV over 4 hours on days 1, 8, and 15 of each 28 day cycle. carfilzomib: Given IV romidepsin: Given IV laboratory biomarker analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Arm A, Cohort 1 (Carfilzomib) | Arm B Cohort 1 (Carfilzomib + Romidepsin) | Arm B Cohort 2 (Carfilzomib + Romidepsin) | Total
Number analyzed (Participants) | 3 | 1 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 1 | 4
  >=65 years | 1 | 0 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 1 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 1 | 1 | 2 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLTs)
Description: To determine the maximum tolerated dose (MTD) by assessing the adverse events experienced by patients of both carfilzomib alone and when taken with romidepsin for dose limiting toxicities (DLT) on days 1 and 15 of the first 28 days of treatment. Toxicities will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v 4.0.
  DLT is defined as any of the following:
  Grade ≥ 2 neuropathy with pain Grade ≥ 3 non-hematologic toxicity Grade ≥ 3 nausea, vomiting, or diarrhea not controlled Grade ≥ 4 fatigue persisting for > 7 days Grade 4 neutropenia (ANC < 500/mm3) occurring for >7 days Febrile neutropenia [ANC < 1000/mm3 with fever Grade ≥ 3 thrombocytopenia persisting for > 7 days Grade ≥ 3 thrombocytopenia associated with bleeding Any toxicity requiring a dose reduction within Cycle 1 Inability to receive Cycle 2, Day 1 dose due to drug related toxicity persisting from Cycle 1 or drug-related toxicity newly encountered on Cycle 2, Day 1
Time Frame: During the first 28 days (1 cycle=28 days) of treatment.
Population: Study terminated early due to slow accrual and not all cohorts enrolled patients. Only number of patients that experienced DLTs are shown below for arms and cohorts that enrolled as data could not be collected regarding MTD
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A, Cohort 1 (Carfilzomib) | Arm B Cohort -1 (Carfilzomib + Romidepsin) | Arm B Cohort 1 (Carfilzomib + Romidepsin
Number analyzed (Participants) | 2 | 1 | 3
Participants | 0 | 0 | 2

2. Secondary Outcome: Overall Response Rate (ORR) of the Disease When Treated With Carfilzomib Alone and When Taken With Romidepsin
Description: Overall Response Rate (ORR) is defined as number of patients who's best response is complete response or partial response. Response will be categorized as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD). The overall response rate of the study treatment will be evaluated based on skin biopsy, CT scans, and blood tests at the beginning of the study as well as every 56 days (2 cycles).
Time Frame: Baseline and every 56 days (2 cycles) while on treatment and up to 4 cycles
Population: Data was not collected for this outcome measure due to study terminating early due to slow accrual.
Arm/Group | Arm A (Carfilzomib) | Arm B (Carfilzomib, Romidepsin)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Duration of Response of the Disease When Treated With Carfilzomib Alone and When Taken With Romidepsin
Description: Duration of response will be defined as the time from the point at which response is achieved until the point of disease progression. The duration of response of the study treatment will be evaluated based on skin biopsy, CT scans, and blood tests at the beginning of the study as well as every 56 days (2 cycles).
Time Frame: Baseline and every 56 days (2 cylces) until disease progression
Population: Data was not collected for this outcome measure due to the study terminating early due to slow accrual.
Arm/Group | Arm A (Carfilzomib) | Arm B (Carfilzomib, Romidepsin)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Progression (TTP) of the Disease When Treated With Carfilzomib Alone and When Taken With Romidepsin
Description: The time to progression (TTP) will be measured as the time from the first dose of study therapy until the point at which disease is determined to have progressed or patients discontinue therapy for toxicity. To measure time to progression, the study treatment will be evaluated based on skin biopsy, CT scans, and blood tests at the beginning of the study as well as every 56 days (2 cycles).
Time Frame: Baseline and every 56 days (2 cycles) until disease progression or toxicity call for discontinuation of treatment
Population: Data was not collected for this outcome measure due to the study terminating early due to slow accrual.
Arm/Group | Arm A (Carfilzomib) | Arm B (Carfilzomib, Romidepsin)
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Proteasome Activity Will be Measured in Peripheral Blood and Tumor Tissue Samples to Observe Proteasome Inhibition While on Treatment
Description: Proteasome inhibition will be measured by evaluating proteasome activity in blood and tumor tissue biopsy specimens while on treatment of carfilzomib alone as well as carfilzomib with romidepsin.
Time Frame: Blood is collected before & after carfilzomib dosing during cycle 1 (days 1, 2, & 8) & cycle 2 (day 1) & Tumor tissue samples obtained at baseline, 1-4 hours post-first dose of carfilzomib (cycle 1 day 1) & 1-4 hours post-carfilzomib on cycle 1 day 8
Population: Data was not collected for this outcome measure due to the study terminating early due to slow accrual.
Arm/Group | Arm A (Carfilzomib) | Arm B (Carfilzomib, Romidepsin)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the study over a 2 and half year period. Adverse events were collected for up to 30 days post 4 cycles ( the most time any patient received treatment on study)
Arm/Group | Arm A, Cohort 1 (Carfilzomib) | Arm B Cohort -1 (Carfilzomib + Romidepsin) | Arm B Cohort 1 (Carfilzomib + Romidepsin
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 2/3
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A, Cohort 1 (Carfilzomib) (N=2) | Arm B Cohort -1 (Carfilzomib + Romidepsin) (N=1) | Arm B Cohort 1 (Carfilzomib + Romidepsin (N=3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A, Cohort 1 (Carfilzomib) (N=2) | Arm B Cohort -1 (Carfilzomib + Romidepsin) (N=1) | Arm B Cohort 1 (Carfilzomib + Romidepsin (N=3)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 2
palpitations (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Edema limbs (General disorders) | 2 | 0 | 1
Edema trunk (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0
Fever (General disorders) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Lymphocyte count increased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 2
Weight loss (Investigations) | 0 | 0 | 1
White blood cell decreased (Investigations) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bronchopulmonary hemorrhage (Metabolism and nutrition disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study terminated early before accrual was met due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes